CLINICAL TRIAL: NCT03212235
Title: Hypofractionated Radiation Therapy Plus Concomitant and Adjuvant Temozolomide for Glioblastoma
Brief Title: Hypofractionated Radiation Therapy for Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Gustavo Nader Marta, Radiation Oncologist and Principal Investigator, Instituto do Cancer do Estado de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypofractionated GBM
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated radiation therapy (Experimental): Hypofractionated radiation therapy Total dose: 60 Gy (20 fractions / 3 Gy per fraction) with concurrent temozolomide 75 mg/m2 given 7 days/week.
  After a 30-days break, adjuvant temozolomide days 1-5 every 28 days for 6 cycles.
  Interventions: Radiation: Hypofractionated radiation therapy

INTERVENTIONS:
Radiation: Hypofractionated radiation therapy — Hypofractionated radiation therapy Total dose: 60 Gy (20 fractions / 3 Gy per fraction)

SUMMARY:
Notwithstanding major improvements in treatment modalities, the prognosis of patients with glioblastoma is poor. Hypofractionated radiation therapy as an alternative of the standard 6-week regimen could be an attractive approach as an effort to prevent tumor cell repopulation and reduction the total treatment period promoting patient comfort and convenience.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 70 years of age with newly diagnosed and histologically confirmed glioblastoma.
* WHO performance status of 2 or less and adequate hematologic, renal, and hepatic function.

Exclusion Criteria:

* Prior diagnosis of cancer, unless disease free for > 3 years
* Previous history of radiotherapy in the head and neck region (except initial larynx tumor - T1, T2 / N0M0).
* Specific severe, active co-morbidities
* Tumor located in the brainstem
* Presence of leptomeningeal carcinomatosis
* Multicentric tumor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  From date of the start of treatment to date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival | 24 months
  The time between the start of treatment and tumor progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto do Cancer do Estado de São Paulo (ICESP) - FMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No